CLINICAL TRIAL: NCT06483815
Title: Comparative Retrospective Analysis of Fungal Positivity Rates During and Post-SARS-CoV-2 Pandemic Periods
Brief Title: Fungal Infections During and After the SARS-CoV-2 Pandemic: A Retrospective Comparison
Status: Enrolling by invitation | Type: Observational
Sponsor: Bekir Sami Uyanık (Other)
Responsible Party: Sponsor-Investigator, Bekir Sami Uyanık, Professor, Hisar Intercontinental Hospital
Organization: Hisar Intercontinental Hospital (Other)
Other Study IDs: ODFUNGAL
Record Dates: First submitted 2024-06-29; First posted 2024-07-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Fungal Infections
Keywords: fungal infections, SARS-CoV-2, pandemic, post-pandemic
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — bronchoalveolar lavage, tracheal aspirate, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The percentages of fungus positivity in the SARS CoV-2 pandemic and SARS CoV-2 post-pandemic period: The study was conducted retrospectively, analyzing a total of 1441 patients. Among these, 623 were during the SARS-CoV-2 pandemic and 818 were in the post-pandemic period. Fungal positivity rates were calculated separately for different fungal agents including Candida species and Aspergillus. These rates were presented as percentages and statistically compared between the two periods.
  Interventions: Diagnostic Test: Culture, İsolation

INTERVENTIONS:
Diagnostic Test: Culture, İsolation — Data on patient demographics, clinical conditions, and fungal infection positivity rates were extracted from hospital records. Fungal positivity rates were calculated based on laboratory results and presented as percentages. Statistical analyses were performed using the Chi-Square test, and p-values were reported.

SUMMARY:
his study aims to retrospectively compare fungal positivity rates between the SARS-CoV-2 pandemic and the post-pandemic periods. During the pandemic, Candida species had a positivity rate of 17.36%, and Aspergillus had a rate of 2.22%. Post-pandemic, these rates decreased to 9.29% and 1.00%, respectively. The overall fungal positivity rate decreased from 9.15% during the pandemic to 5.13% post-pandemic. Statistical analysis revealed a significant decrease in fungal positivity rates post-pandemic (p < 0.01). These findings underscore the effectiveness of post-pandemic healthcare interventions and infection control strategies.

DETAILED DESCRIPTION:
The study aims to retrospectively compare fungal positivity rates by focusing on Candida and Aspergillus species during the SARS-CoV-2 pandemic and in the post-pandemic period. The dataset includes samples collected during the pandemic period (N=623) and the subsequent post-pandemic period (N=818). Fungal positivity rates were calculated and statistically analyzed using chi-square tests, and significance was determined as p<0.01.

During the SARS-CoV-2 pandemic, Candida species showed a positivity rate of 17.36%, while the rate in the post-pandemic period significantly decreased to 9.29% (p=0.002). In contrast, Aspergillus species did not show a significant change in positivity rates between the pandemic (2.22%) and post-pandemic (1.00%) periods (p=0.186, NS).

Overall, the study provides valuable insights into the epidemiology of fungal infections during and after the SARS-CoV-2 pandemic, suggesting possible shifts in fungal pathogen prevalence and healthcare priorities. The findings contribute to the development of targeted healthcare strategies and surveillance measures for fungal infections in the post-pandemic era.

Study Design: Retrospective comparative analysis

Data Analysis: Chi-square tests, p<0.01 considered significant

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age of both genders

Exclusion Criteria:

* Patients under 18 years of age,
* Patients whose demographic, clinical and laboratory data investigated in the study could not be accessed, patients who were diagnosed with fungal infection during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pneumonia according to clinical, laboratory and radiological data in the chest diseases, infectious diseases and intensive care unit of Hisar HIntercontinental Hospital
Sampling Method: Probability Sample
Enrollment: 1441 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Fungal positivity rates during the SARS-CoV-2 pandemic period and post-pandemic period | 2020-2024
  Fungal infection data from samples of patients, 623 of whom were during the SARS-CoV-2 epidemic and 818 of whom were in the post-epidemic period, were retrospectively examined. Fungal positivity rates for different fungal agents such as Candida species and Aspergillus were calculated separately and compared statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Gözüküçük, Study Director — Hisar Hospital Responsible Manager
Locations (1):
- Hisar Hospital Intercontinental, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No